CLINICAL TRIAL: NCT06619249
Title: Effect of Endurance Training-Induced Coenzyme Q10 (CoQ10) Supplementation on Myokine, Exerkine Secretion and Cognitive Functions in Long-Distance Runners
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AWFiS/2024_3_ZJ
Record Dates: First submitted 2024-08-06; First posted 2024-10-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-08

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Coenzyme Q10; Supplementation; Myokine; Exerkine; Cognition; Long-distance runners
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CoQ10-treated participants (Experimental): The participants will be treated with CoQ10 supplements
  Interventions: Dietary Supplement: CoQ10 supplementation
- Placebo-treated participants (Placebo Comparator): The participants will be treated with placebo
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: CoQ10 supplementation — Long-distance runners will be supplemented with CoQ10 for 4 weeks in cross-over manner with 4 weeks of wash out period.
  Arms: CoQ10-treated participants
Dietary Supplement: Placebo supplementation — Long-distance runners will be supplemented with placebo for 4 weeks in cross-over manner with 4 weeks of wash out period.
  Arms: Placebo-treated participants

SUMMARY:
The goal of this clinical trial is to learn if CoQ10 amplifies endurance training-induced myokine and exerkine secretion and if those changes influences cognition in long-distance runners.

Does 4-week high-dosage CoQ10 supplementation increase the secretion of myokine, exerkine sercetion? Does the above-mentioned intervention improve the cognitive function in long distance runners?

Participants will:

Take CoQ10 or a placebo every day for 4 weeks. Visit the laboratory once every 4 weeks for checkups and tests. Keep the participants' food and training diary.

ELIGIBILITY:
Inclusion Criteria:

* training experienced for minimum 2 years
* running training at least 2 times per week
* Personal Best on 10k (<50 minutes)

Exclusion Criteria:

* taking supplements which can interrupt primary outcomes (vitamin D, omega-3 fatty acids)
* injured in last 6 months to avoid n number reduction

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive funtions as a result of CoQ10 supplementation measured via cogntitive function test. | The investigators are going to check this hypothesis after 4 weeks of high-dose supplementation with CoQ10
  The investigators assume that supplementation with CoQ10 will change cognition (measured via cognitive function tests - Stroop Test, Trial Making Test A and Trial Making Test B) in long-distance runners. The results will be obtained as time (seconds) needed to complete tasks while testing.
Change in myokine and exerkine concentration in the blood plasma as a result of CoQ10 supplementation. | The investigators are going to check this hypothesis after 4 weeks of high-dose supplementation with CoQ10
  The investigators will assess the concentration of blood myokine and exerkine concentration (pg or ug/dl) of blood plasma using the colorimetric method.

SECONDARY OUTCOMES:
Change in aerobic capacity measured via direct test to volitional exhaustion on a motorized treadmill | The investigators are going to check this hypothesis after 4 weeks of high-dose supplementation with CoQ10
  The investigators assume that supplementation with CoQ10 will change the aerobic capacity (oxygen uptake in ml-1 x min-1 x kg-1) in long-distance runners. The determination of aerobic capacity will be done through progressive test to volitional exhaustion on a motorized treadmill and gas analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland